CLINICAL TRIAL: NCT05911373
Title: Serratus Plane Block Versus Serratus Plane Block Plus Parasternal Block on Postoperative Opioid Consumption and Dermatomal Analyses for Breast Surgery
Brief Title: Serratus Plane Block Versus Serratus Plane Block Plus Parasternal Block Combination for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ataunibreastanalgesia
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Analgesia; Cancer, Breast
MeSH Terms: conditions — Agnosia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group serratus (Placebo Comparator): preoperative superficial serratus block with local anaesthetics and parasternal block with saline
  Interventions: Other: group serratus plan block
- group serratus and parasternal (Active Comparator): preoperative superficial serratus block and parasternal block with local anaesthetics
  Interventions: Other: group serratus and parasternal plan block

INTERVENTIONS:
Other: group serratus plan block — preoperativelly, Superficial Serratus Block performed with 30 ml %0.25 Bupivacaine and Parasternal Block performed with 10 ml saline
  Arms: group serratus
Other: group serratus and parasternal plan block — preoperativelly, Superficial Serratus Block performed with 30 ml %0.25 Bupivacaine and Parasternal Block performed with 10 ml %0.25 Bupivacaine
  Arms: group serratus and parasternal

SUMMARY:
Mastectomy is a technique often used in breast cancer surgery. Patients experience moderate to severe pain postoperatively after this procedure. Various plane blocks, NSAIDs, and opioid analgesics can be administered to these patients as components of multimodal analgesia. In the the study, the investigators aimed to evaluate the analgesic effects of the serratus plane block, the parasternal block added to the serratus plane block, and the dermatomal differences.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologist's physiologic state I-III patients
2. To undergo Mastectomy Surgery
3. Being between the ages of 18-65 years

Exclusion Criteria:

* Having a known heart, kidney, liver or hematological disease
* Having a history of peptic ulcer, gastrointestinal bleeding, allergy, chronic pain
* Routine analgesic use and history of analgesic use in the last 24 hours
* Not willing to participate in the study
* Uncooperative patients who have coagulopathy or use anticoagulant drugs
* To be allergic to one of the drugs to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | First 24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (between 0-10; 0: no pain, 10:worst pain) score
Sensory Assessment | 24 hours
  Sensory Assessment will be performed on patients following the block procedure with pinprick test.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsnü Kürşad, Study Director — Ataturk University
Locations (1):
- Ali Ahiskalioglu, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Hu NQ, He QQ, Qian L, Zhu JH. Efficacy of Ultrasound-Guided Serratus Anterior Plane Block for Postoperative Analgesia in Patients Undergoing Breast Surgery: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Pain Res Manag. 2021 Oct 25;2021:7849623. doi: 10.1155/2021/7849623. eCollection 2021. PMID 34733377
- [Background] Piraccini E, Biondi G, Corso RM, Maitan S. The use of rhomboid intercostal block, parasternal block and erector spinae plane block for breast surgery. J Clin Anesth. 2020 Feb;59:10. doi: 10.1016/j.jclinane.2019.06.004. Epub 2019 Jun 6. No abstract available. PMID 31176954